CLINICAL TRIAL: NCT06407375
Title: Assessment of Renal Function by Multiparametric MRI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: mpMRI Kidney
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mpMRI — mpMRI

SUMMARY:
Metabolic syndrome is a collection of conditions that affect at least three of the following five criteria: abdominal obesity, high blood pressure, high fasting glucose levels, high triglyceride levels, and low levels of high-density lipoprotein (HDL) cholesterol. Chronic kidney disease (CKD) is a common complication of metabolic syndrome, with an estimated prevalence of 13-40%. Early diagnosis of progressive conditions before the onset of reduced glomerular filtration rate (GFR) or albuminuria may be of clinical benefit but is not possible at present. Furthermore, the diagnosis and quantification of CKD in the context of metabolic syndrome is challenging due to the lack of reliable diagnostic biomarkers, and the current methods may not accurately reflect kidney function in patients with metabolic syndrome. Magnetic resonance imaging (MRI) has been sparsely explored as a potential tool to assess renal perfusion, oxygenation, and fibrosis. Multiparametric MRI (mpMRI) combines several different imaging techniques to provide a more comprehensive evaluation of tissue structure and function. These techniques hold promise for non-invasive assessment of kidney function, but their clinical utility is still largely experimental. Therefore, we aim to conduct an exploratory study to investigate the reliability, reproducibility as well as the validity of parameters for kidney function of multiparametric MRI as well as compare these parameters in between healthy patients and patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed metabolic syndrome

Exclusion Criteria:

* MRI exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: Healthy participants of different age groups
Period: Overall Study
Arm/Group | Healthy Participants
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Participants
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Serum Creatinine [Mean (Standard Deviation); unit: µmol/L] — Serum Creatinine (measured prior to MRI)
  µmol/L | 72 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: T1 Time
Description: T1 relaxation time (MR characteristic of the human tissue, measured in ms)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Healthy participants: Healthy participants
Arm/Group | Healthy participants
Number analyzed (Participants) | 46
ms | 1500 (15)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT06407375/Prot_SAP_000.pdf